CLINICAL TRIAL: NCT03536702
Title: Effect of Group Led Creative Writing on Mood in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Monika Joshi, Assistant Professor, Department of Medicine, Division of Hematology-Oncology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PSCI 18-005
Record Dates: First submitted 2018-03-28; First posted 2018-05-25 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Cancer Patients

STUDY DESIGN:
Intervention Model Description: Participants will be randomized within strata formed by cancer type in order to assure that these potentially important confounding variables are balanced across groups. Patients will be enrolled on a rolling basis over a three-month period, allowing patients in intervention arm to participate in 3 months workshops (workshops would be held once every 2 weeks). Patients in control arm will be provided a book (Writing Down Bones by Natalie Goldberg) about creative writing and will be asked to do activities for 1.5 hours every 2 weeks. After three months, control group participants can join creative writing workshops at their discretion for the remaining period for writing workshops. Both group members will receive follow up surveys twice a month for two months at the completion of the participant's three-month study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Writing Workshop (Experimental): The intervention arm will receive a dedicated workshop for one and a half hours every 2 weeks for 3 months.
  Interventions: Other: Creative Writing Workshop
- Independent Writing - Control Group (Active Comparator): The control arm will receive a book (i.e., Writing Down Bones by Natalie Goldberg) on creative writing and asked to read and do writing activities for one and a half hours once every two weeks for 3 months.
  Interventions: Other: Independent Writing - Control Group

INTERVENTIONS:
Other: Creative Writing Workshop — This group will participate in a writing workshop in group sessions.
  Arms: Creative Writing Workshop
Other: Independent Writing - Control Group — This group will receive a book for a self writing session.
  Arms: Independent Writing - Control Group

SUMMARY:
The primary purpose of this study is to determine whether creative writing in newly diagnosed cancer patients and those with recent progression in their disease will have a positive impact on their mental health. Using a randomized controlled trial approach, emotion thermometers will be employed to evaluate participants' responses on a number of domains, such as anxiety, depression, despair, and anger along with a series of survey questions to monitor changes in depressive and anxiety symptoms. Open-ended survey questions will be used to capture how a creative writing intervention impacts participants' experience of their illness. Melissa Greene's Write from the Heart program focuses more on creative writing rather than cancer focused topics. Patients in the intervention arm will complete -one and a half hour group sessions every two weeks over the span of 3 months. Participants in the active control arm will be provided a book (i.e., Writing Down Bones by Natalie Goldberg) about creative writing and will be asked to do activities for 1.5 hrs every 2 weeks for a period of 3 months.

DETAILED DESCRIPTION:
Mental wellness before and after intervention in both arms. A validated Emotional Thermometer Scales will be used to predict changes in parameters reflecting participants' mental health pre- and post-intervention. Survey questions focused on symptoms of depression and anxiety will be used to monitor for changes in mental wellness pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed with any stage or type of cancer within 3 months OR progression of disease within 3 months of enrollment. Recurrence of cancer within 3 months of enrollment would also be eligible as it will be considered as progression of cancer Ability to understand English language and ability to write without any functional difficulty ECOG performance status 0-3

Exclusion Criteria:

Inability to give informed consent Severe psychiatry illness (e.g., uncontrolled depression, schizophrenia or psychosis) Severe cognitive impairment Pregnant females Inability to write or understand English

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, MD, Principal Investigator — Penn State Hershey Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DOI: 10.1200/JCO.2017.35.31_suppl.178 Journal of Clinical Oncology 35, no. 31_suppl (November 2017) 178-178.
- See also: Abstract presented at Palliative Care Symposium 11/2017 — http://ascopubs.org/doi/abs/10.1200/JCO.2017.35.31_suppl.178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 subjects signed consent. Results reported are for completers only. Completers are participants who signed consent, were randomized, completed baseline measures and took at least one class after baseline.
Period: Overall Study
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Started | 40 | 20
Completed (Competers are those who signed consent took baseline measures and at least one class) | 26 | 8
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Population: Following the Intention-to-treat (ITT) principle, we report the status of all the 60 consented participants, who have been randomized with 1:2 ratio to two groups (control and intervention). Of those 60, 34 completed the baseline measures and took one class.
Groups:
- Total: Total of all reporting groups
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group | Total
Number analyzed (Participants) | 26 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.8) | 57.8 (10.1) | 61.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 4 | 22
  Male | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 25 | 7 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mood Score Baseline Emotional Thermometer Scale subscale 1-distress [Median (Full Range); unit: units on a scale] — Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.
  units on a scale | 2 [0 to 6.5] | 2 [0 to 5] | 2 [0 to 6.5]
Emotional Thermometer subscale 2- anxiety baseline [Median (Full Range); unit: units on a scale] — Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.
  units on a scale | 4 [0 to 10] | 5.5 [1 to 8] | 4 [0 to 10]
Emotional Thermometer subscale 3- depression baseline [Median (Full Range); unit: units on a scale] — Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score..
  units on a scale | 1 [0 to 9] | 3 [0 to 8] | 1.2 [0 to 9]
Emotional Thermometer subscale 4- anger baseline [Median (Full Range); unit: units on a scale] — Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.
  units on a scale | 0.2 [0 to 7] | 2.5 [0 to 10] | 0.5 [0 to 10]
Emotional Thermometer subscale 5- need help baseline [Median (Full Range); unit: units on a scale] — Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.
  units on a scale | 1 [0 to 7] | 1.5 [0 to 8] | 1 [0 to 8]
Emotional Thermometer score (total) at baseline [Median (Full Range); unit: units on a scale] — A validated Emotional Thermometer Scales will be used to predict changes in parameters pre and post-intervention. The validated Emotional Thermometer Scale (ETS) has five dimensions (distress, anxiety, depression, anger and need help), which are all continuous variables and range from 0 (best) to 10 (worst). Both the individual scores will be analyzed for each dimension as well as a sum of the five scores will be collected to represent average mood score.
  units on a scale | 2 [0 to 25] | 9.5 [2 to 21] | 3 [0 to 25]
Self Reported Somatic Symptoms baseline [Median (Full Range); unit: units on a scale] — Self-reported somatic symptoms pre and post intervention in two groups. We will use the Somatic Symptom Scale - 8 (SSS-8) to quantify somatic symptom burden. The scale is composed of 8 questions with options to choose a score of 0 (not at all) - 4 (very much) to describe degree of distress caused by individual somatic symptoms. A total of the 8 scores is used as a final value for the SSS-8, with higher scores indicating worse Somatic Symptom severity
  units on a scale | 7 [0 to 18] | 7 [2 to 16] | 7 [0 to 18]
Depression Symptoms baseline [Median (Full Range); unit: units on a scale] — Severity of depression symptoms before and after intervention between two groups. The validated depression questionnaire, the Patient Health Questionnaire-9 (PHQ-9), will be used to predict changes. This questionnaire includes 9 questions, that describes individual symptoms of depression and asks individuals to asses how much each depression symptoms has bothered them in the last two weeks, from 0 (not at all) to 3 (nearly every day). The total score is compiled to represent a final depression severity score, with higher scores indicating worse severity, at a maximum value of 27 points
  units on a scale | 3 [0 to 13] | 4 [2 to 8] | 3 [0 to 13]
Anxiety Symptoms baseline [Median (Full Range); unit: units on a scale] — The validated anxiety questionnaire, the Generalized Anxiety Disorder - 7 Scale, will be used to predict changes. This includes 7 questions describing symptoms of generalized anxiety, asking individual patients to rate how much those symptoms have bothered the individual in the past two weeks, from a score of 0 (not at all) to 3 (nearly every day). The total of the scores will be used to represent anxiety symptoms score, with a minimum score of 0 and a maximum score of 21, with higher score representing increasing severity of anxiety
  units on a scale | 3 [0 to 12] | 3 [0 to 9] | 3 [0 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Emotional Thermometer Subscale 1- Distress at Final
Description: Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 0 [0 to 4] | 1.5 [0 to 4.5]

2. Primary Outcome: Emotional Thermometer Subscale 2 - Anxiety at Final
Description: as for outcome 1
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 1 [0 to 6] | 2.5 [1 to 7]

3. Primary Outcome: Emotional Thermometer Subscale 3 - Depression at Final
Description: Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.re.
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 0 [0 to 6] | 2 [0 to 7]

4. Primary Outcome: Emotional Thermometer Subscale 4-anger at Final
Description: as for outcome 1
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 0 [0 to 4] | 1.5 [0 to 5]

5. Primary Outcome: Emotional Thermometer Subscale 5-need Help at Final
Description: as for outcome 1
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 0 [0 to 6] | 0.5 [0 to 3]

6. Primary Outcome: Emotional Thermometer Score (Total) at Final
Description: Mood scores before and after intervention (after completion of entire session this may vary as some patients may not be able to complete six sessions). A validated Emotional Thermometer Scales (ETS) will be used to predict changes pre and post-intervention. The validated ETS has five dimensions (distress, anxiety, depression,anger, need help), which are all continuous variables and range from 0 to 10 with 0 being no emotional symptoms and 10 extremely emotional. Individual scores will be analyzed as well as a sum of the five scores will be collected to represent average mood score.score.
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
units on a scale | 2 [0 to 25] | 9.5 [2 to 21]

7. Secondary Outcome: Depression Symptoms
Description: Severity of depression symptoms before and after intervention between two groups. The validated depression questionnaire, the Patient Health Questionnaire-9 (PHQ-9), will be used to predict changes. This questionnaire includes 9 questions, that describes individual symptoms of depression and asks individuals to asses how much each depression symptoms has bothered them in the last two weeks, from 0 (not at all) to 3 (nearly every day). The total score is compiled to represent a final depression severity score, with higher scores indicating worse severity, at a maximum value of 27 points.
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 21 | 5
units on a scale | 3 [0 to 18] | 3 [1 to 16]

8. Secondary Outcome: Anxiety Symptoms
Description: Severity of anxiety symptoms before and after intervention between two groups. The validated anxiety questionnaire, the Generalized Anxiety Disorder - 7 Scale, will be used to predict changes. This includes 7 questions describing symptoms of generalized anxiety, asking individual patients to rate how much those symptoms have bothered the individual in the past two weeks, from a score of 0 (not at all) to 3 (nearly every day). The total of the scores will be used to represent anxiety symptoms score, with a minimum score of 0 and a maximum score of 21, with higher score representing increasing severity of anxiety.
Time Frame: 4 months
Reporting Status: Not Posted

9. Secondary Outcome: Self Reported Somatic Symptoms at Final
Description: Self-reported somatic symptoms pre and post intervention in two groups. We will use the Somatic Symptom Scale - 8 (SSS-8) to quantify somatic symptom burden. The scale is composed of 8 questions with options to choose a score of 0 (not at all) - 4 (very much) to describe degree of distress caused by individual somatic symptoms. A total of the 8 scores is used as a final value for the SSS-8, with higher scores indicating worse Somatic Symptom severity.
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 22 | 5
units on a scale | 7 [1 to 16] | 5 [1 to 20]

10. Secondary Outcome: Depression Symptoms at Final
Description: as for outcome 7
Time Frame: 4 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 21 | 5
units on a scale | 3 [0 to 18] | 3 [1 to 16]

11. Other Pre Specified Outcome: Status of Cancer at Consent
Description: Comparison of status of cancer (stable, progressing, in remission) between intervention and control group.
Time Frame: consent
Measure: Count of Participants; unit: Participants
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
Participants
  Cured | 2 | 1
  New | 10 | 2
  Progression | 5 | 0
  Stable | 9 | 5

12. Other Pre Specified Outcome: Number of Subjects Who Were Admitted to the Hospital and ER Admissions During Study Time
Description: Difference in number of emergency room visits and hospitalizations during study period between control and intervention group
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
Participants | 5 | 0

13. Other Pre Specified Outcome: Number of Subject That Were Not Hospital or ER Admissions After Study
Description: as for outcome 12
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
Participants | 20 | 4

14. Other Pre Specified Outcome: Number of Emergency Room Visits and Hospitalizations Per Subject
Description: Difference in number of emergency room visits and hospitalizations per subject during study period between control and intervention group
Time Frame: 4 months
Measure: Number; unit: ER visits and hospitalizations
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
ER visits and hospitalizations | 6 | 4

15. Other Pre Specified Outcome: Status of Cancer at End of Study
Description: Comparison of status of cancer (stable, progressing, in remission) between intervention and control group.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
Participants
  stable | 18 | 5
  Progression | 8 | 3

16. Other Pre Specified Outcome: Number of Subject That Were Not Hospitalized or in the Emergency Room During Study Time
Description: Difference in number of emergency room visits and hospitalizations by subject during study period between control and intervention group
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
Number analyzed (Participants) | 26 | 8
Participants | 21 | 8

ADVERSE EVENTS:
Time Frame: up to 4 months
Arm/Group | Creative Writing Workshop | Independent Writing - Control Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/8
Other Adverse Events (participants affected / at risk) | 0/26 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT03536702/Prot_SAP_000.pdf